CLINICAL TRIAL: NCT01571453
Title: Randomised, Double-blind, Parallel-group, Active-comparator (Venlafaxine Extended Release), Fixed-dose Study of [Vortioxetine] Lu AA21004 in Major Depressive Disorder in Asian Countries
Brief Title: Study of Vortioxetine (Lu AA21004) in Major Depressive Disorder in Asian Countries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13926A
Record Dates: First submitted 2012-03-28; First posted 2012-04-05 (Estimated); Results first posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Major Depressive Disorder
Keywords: MDD
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vortioxetine (Lu AA21004) (Experimental)
  Interventions: Drug: Vortioxetine (Lu AA21004)
- Venlafaxine extended release (Active Comparator)
  Interventions: Drug: Venlafaxine extended release

INTERVENTIONS:
Drug: Vortioxetine (Lu AA21004) — 10 mg/day
  Other Names: Brintellix
  Arms: Vortioxetine (Lu AA21004)
Drug: Venlafaxine extended release — 150 mg/day
  Other Names: Efexor® XL
  Arms: Venlafaxine extended release

SUMMARY:
This study will be conducted with the aim of investigating the efficacy, safety and tolerability of 10 mg/day Vortioxetine in Asian patients compared to an approved active comparator (venlafaxine extended release 150 mg/day).

ELIGIBILITY:
Inclusion Criteria:

* The patient suffers from recurrent MDD as the primary diagnosis according to DSM-IVTR™ criteria. The current Major Depressive Episode (MDE) should be confirmed using the Mini International Neuropsychiatric Interview (MINI)
* The patient has a MADRS total score ≥26
* The patient has a CGI-S score ≥4
* The reported duration of the current MDE is ≥3 months.

Other inclusion criteria may apply.

Exclusion Criteria:

- The patient meets any of the exclusion criteria listed in the protocol or, in the investigator's opinion, is unlikely to comply with the protocol or is unsuitable for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

REFERENCES:
- [Derived] Wang G, Zhao K, Reynaud-Mougin C, Loft H, Ren H, Eriksen HF, Ettrup A. Successfully treated patients with vortioxetine versus venlafaxine: a simplified cost-effectiveness analysis based on a head-to-head study in Asian patients with major depressive disorder. Curr Med Res Opin. 2020 May;36(5):875-882. doi: 10.1080/03007995.2020.1723072. Epub 2020 Feb 13. PMID 31990207
- [Derived] Wang G, Gislum M, Filippov G, Montgomery S. Comparison of vortioxetine versus venlafaxine XR in adults in Asia with major depressive disorder: a randomized, double-blind study. Curr Med Res Opin. 2015 Apr;31(4):785-94. doi: 10.1185/03007995.2015.1014028. Epub 2015 Feb 19. PMID 25650503

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In- or outpatients with a primary diagnosis of recurrent of Major Depressive Disorder (MDD) were recruited for this study from China, South Korea, Taiwan, and Thailand.
Pre-assignment Details: A Screening Visit was held approximately 7 days prior to group assignment (group assignment was held during the Baseline Visit). Patients who met each of the inclusion criteria at the Screening and Baseline Visits and none of the exclusion criteria at the Screening and/or Baseline Visit were eligible to participate in this study.
Groups:
- Vortioxetine: Vortioxetine (Lu AA21004): 10 mg/day
- Venlafaxine: Venlafaxine extended release 150 mg/day
Period: Overall Study
Arm/Group | Vortioxetine | Venlafaxine
Started | 211 | 226
Completed | 173 | 164
Not Completed | 38 | 62
Not completed — Adverse Event | 14 | 32
Not completed — Lack of Efficacy | 8 | 3
Not completed — Non-compliance | 2 | 4
Not completed — Protocol Violation | 1 | 5
Not completed — Withdrawal of consent | 5 | 13
Not completed — Lost to Follow-up | 4 | 2
Not completed — Administrative or other reason(s) | 4 | 3

BASELINE CHARACTERISTICS:
Population: The all-patients-treated set (APTS) comprises all randomized patients who took at least one dose of IMP.
  Baseline age and gender is based on the APTS. Baseline efficacy outcome measures is based on the full-analysis set (FAS).
Groups:
- Venlafaxine: Venlafaxine extended release: 150 mg/day
- Total: Total of all reporting groups
Arm/Group | Vortioxetine | Venlafaxine | Total
Number analyzed (Participants) | 211 | 226 | 437
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (12.4) | 40.7 (12.3) | 40.1 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 139 | 262
  Male | 88 | 87 | 175
MADRS total score [Mean (Standard Deviation); unit: units on a scale] — Montgomery and Asberg Depression Rating Scale (MADRS) is a ten-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). Definitions of severity are provided at two-point intervals. The total score of the ten items ranges from 0 to 60. The higher the score, the more severe.
  units on a scale | 32.3 (4.6) | 32.3 (4.5) | 32.3 (4.6)
HAM-A total score [Mean (Standard Deviation); unit: units on a scale] — Hamilton Anxiety Rating Scale (HAM-A) is a 14-item rating scale designed to assess the global anxiety. Each symptom is rated from 0 (absent) to 4 (maximum severity). The total score of the 14 items ranges from 0 to 56. Total score from 0 to 56; higher score indicates greater anxiety.
  units on a scale | 20.6 (7.3) | 21.1 (7.0) | 20.9 (7.1)
CGI-S score [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impression Scale - Severity of Illness (CGI-S) provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients). Higher score indicates that the patient is more ill.
  units on a scale | 4.8 (0.7) | 4.9 (0.7) | 4.9 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in MADRS Total Score at Week 8
Description: Montgomery and Asberg Depression Rating Scale (MADRS) is a ten-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). Definitions of severity are provided at two-point intervals. The total score of the ten items ranges from 0 to 60. The higher the score, the more severe, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Baseline and Week 8
Population: The full-analysis set (FAS) comprises all patients in the APTS who had a valid baseline assessment and at least one valid post-baseline assessment of the MADRS total score.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine | Venlafaxine
Number analyzed (Participants) | 209 | 215
units on a scale | -19.36 (0.70) | -18.16 (0.68)
Statistical Analysis 1: Comparison: Vortioxetine vs Venlafaxine; The sample size calculation was based on a non-inferiority comparison of the treatment groups in the change from baseline to Week 8 in MADRS total score using a two-sided 95% CI against a margin of +2.5 points. Assuming a standard deviation of 9.0 points and an expected true mean difference between treatments of 0 points, a total of 410 patients (205 per treatment group) were needed to provide a power of 80% for correctly concluding non-inferiority; Test type: Non-Inferiority or Equivalence — Vortioxetine was declared to be non-inferior to venlafaxine if the upper limit of the calculated two-sided 95% confidence interval for the treatment difference at Week 8 between vortioxetine and venlafaxine was less than +2.5 MADRS units versus venlafaxine; p = 0.199, ANCOVA — No adjustments for multiple comparisons were made; LOCF was used; Mean Difference (Final Values) = -1.20, 95% CI [-3.03 to 0.63], Standard Error of Mean 0.93

2. Secondary Outcome: Change in CGI-S Score From Baseline to Week 8
Description: Clinical Global Impression Scale - Severity of Illness (CGI-S) provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients). Higher score indicates that the subject is more ill, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine | Venlafaxine
Number analyzed (Participants) | 209 | 215
units on a scale | -2.26 (0.09) | -2.12 (0.09)
Statistical Analysis 1: Comparison: Vortioxetine vs Venlafaxine; The same ANCOVA methodology as for the primary endpoint was used; Test type: Superiority or Other; p = 0.228, ANCOVA — No adjustments for multiple comparisons were made; LOCF was used; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.39 to 0.09], Standard Error of Mean 0.12

3. Secondary Outcome: CGI-I Score at Week 8
Description: The Clinical Global Impression - Global Improvement (CGI-I) provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). In all cases, the assessment should be made independent of whether the rater believes the improvement is drug-related or not. Higher score = more affected.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine | Venlafaxine
Number analyzed (Participants) | 209 | 215
units on a scale | 1.99 (0.08) | 2.14 (0.08)
Statistical Analysis 1: Comparison: Vortioxetine vs Venlafaxine; The same ANCOVA methodology as for the primary endpoint was used; Test type: Superiority or Other; p = 0.174, ANCOVA — No adjustments for multiple comparisons were made; LOCF was used; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.35 to 0.06], Standard Error of Mean 0.11

4. Secondary Outcome: Change in HAM-A Total Score From Baseline to Week 8
Description: Hamilton Anxiety Rating Scale (HAM-A) is a 14-item rating scale designed to assess the global anxiety. Each symptom is rated from 0 (absent) to 4 (maximum severity). The total score of the 14 items ranges from 0 to 56. Higher score indicates greater anxiety, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine | Venlafaxine
Number analyzed (Participants) | 209 | 215
units on a scale | -11.38 (0.48) | -10.56 (0.47)
Statistical Analysis 1: Comparison: Vortioxetine vs Venlafaxine; The same ANCOVA methodology as for the primary endpoint was used; Test type: Superiority or Other; p = 0.207, ANCOVA — No adjustments for multiple comparisons were made; LOCF was used; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-2.09 to 0.45], Standard Error of Mean 0.65

5. Secondary Outcome: MADRS Response at Week 8 (Response Defined as a ≥50% Decrease in the MADRS Total Score From Baseline)
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Vortioxetine | Venlafaxine
Number analyzed (Participants) | 209 | 215
percentage of patients | 66.5 | 61.4
Statistical Analysis 1: Comparison: Vortioxetine vs Venlafaxine; Test type: Superiority or Other; p = 0.272, Regression, Logistic — Wald's Test. No adjustments for multiple comparisons were made; Odds Ratio (OR) = 1.25, 95% CI [0.84 to 1.86]

6. Secondary Outcome: Remission at Week 8 (Remission Defined as a MADRS Total Score ≤10)
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Vortioxetine | Venlafaxine
Number analyzed (Participants) | 209 | 215
percentage of patients | 43.1 | 41.4
Statistical Analysis 1: Comparison: Vortioxetine vs Venlafaxine; Test type: Superiority or Other; p = 0.731, Regression, Logistic — Wald's Test. No adjustments for multiple comparisons were made; Odds Ratio (OR) = 1.07, 95% CI [0.73 to 1.58]

7. Secondary Outcome: Number of Adverse Events
Time Frame: Baseline to Week 12

ADVERSE EVENTS:
Time Frame: Baseline to 12 weeks
Arm/Group | Vortioxetine | Venlafaxine
Serious Adverse Events (participants affected / at risk) | 2/211 | 8/226
Other Adverse Events (participants affected / at risk) | 90/211 | 124/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine (N=211) | Venlafaxine (N=226)
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 2
Varicocele (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine (N=211) | Venlafaxine (N=226)
Constipation (Gastrointestinal disorders) | 9 | 18
Dry mouth (Gastrointestinal disorders) | 12 | 24
Dyspepsia (Gastrointestinal disorders) | 11 | 9
Nausea (Gastrointestinal disorders) | 51 | 53
Accidental overdose (Injury, poisoning and procedural complications) | 10 | 12
Decreased appetite (Metabolism and nutrition disorders) | 10 | 23
Dizziness (Nervous system disorders) | 18 | 32
Headache (Nervous system disorders) | 17 | 16
Insomnia (Psychiatric disorders) | 5 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No